CLINICAL TRIAL: NCT00004226
Title: Phase I/II Study of High Dose Limited Volume Postoperative Reirradiation in Recurrent or Second Primary Carcinoma of the Head and Neck
Brief Title: Radiation Therapy Following Surgery in Treating Patients With Recurrent or Second Primary Cancer of the Head and Neck Following Previous Radiation Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067467; UAB-RAD-9601; UAB-F970430006; NCI-G99-1656
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2004-07

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent metastatic squamous neck cancer with occult primary
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of radiation therapy following surgery in treating patients who have recurrent or second primary cancer of the head and neck following previous radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the survival and local control in previously irradiated patients at high risk for local failure following regional resection of recurrent or second primary head and neck cancer.
* Determine the acute and late toxicities of this treatment in these patients.
* Determine the pattern of disease failure in these patients on this treatment.
* Determine any change in quality of life in these patients on this treatment.

OUTLINE: Patients receive fractionated doses of radiotherapy five times weekly for 6 weeks.

Quality of life is assessed prior to study, 2 months after radiotherapy, every 3 months for remainder of year 1, every 4 months for years 2-3, every 6 months for years 4-5, and then annually thereafter.

Patients are followed 2 months after radiotherapy, every 3 months for year 1, every 4 months for year 2, every 6 months for years 3-5, and then annually thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the mucosa, recurrent (primary and/or nodal), or a second primary (positive or negative nodal), of one of the following:

  * Oral cavity
  * Oropharynx
  * Hypopharynx
  * Larynx
  * Paranasal sinus
  * Neck disease of unknown origin
* No distant metastases
* No primary in the nasopharynx
* Must have complete gross resection of disease
* Must have positive final margins, soft tissue extension of primary, positive extracapsular extension of lymph node disease, or at least 4 positive nodes without extracapsular extension
* Reirradiation field must overlap the previous field for a minimum of 3 cm in height, width, and length

  * At least 6 months since prior radiotherapy with an overlap volume of at least 45 Gy
* No grade 3 or 4 toxicity for the following organ tissues:

  * RTOG grade 3 or 4 skin, subcutaneous tissue, larynx, joint, or RTOG grade 4 mucous membrane or bone from prior radiotherapy
* Radiotherapy must begin within 6-12 weeks of surgery
* Prior radiotherapy records must be available

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant
* No history of invasive malignancy that would be expected to cause death within 3 years

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: James L. Pearlman, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (3):
- United States (3):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida